CLINICAL TRIAL: NCT04280445
Title: Acceptance and Commitment Therapy for Older Adults Experiencing Psychological Distress: A Hermeneutic Single Case Efficacy Design (HSCED) Series
Brief Title: Acceptance and Commitment Therapy for Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lincoln (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 191201
Record Dates: First submitted 2020-02-19; First posted 2020-02-21 (Actual); Results first posted 2021-11-02 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2020-01

CONDITIONS: Psychological Distress; Anxiety; Depression
Keywords: Aging; Acceptance and Commitment Therapy; Psychological distress; Anxiety; Depression; Hermeneutics
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Intervention Model Description: The study will employ an adjudicated Hermeneutic Single Case Efficacy Design (HSCED) series with three participants. Following Elliott's (2002; Elliott et al., 2009) approach, a crucial aspect of HSCED research is the formation of rich case records. Developed for each client, these consist of data from various time points in the study, and include demographic, quantitative (outcome measures, treatment fidelity measures etc.) and qualitative sources (Change Interview, therapy feedback, therapy process notes and recordings). The rich case records are then cross-referenced and synthesised into an affirmative and sceptic brief. These briefs are then presented to an expert panel to be adjudicated on the process of change. The resulting decisions will then allow for a between-participant analysis of what components contributed towards change and why.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Psychological therapy (Experimental): All participants will receive psychological therapy. There will be no placebos or waiting list controlled participants to compare findings to.
  Interventions: Other: Psychological therapy

INTERVENTIONS:
Other: Psychological therapy — Acceptance and Commitment Therapy (ACT) is a trans-diagnostic approach which aims to promote better living by supporting clients through six key processes (e.g. mindfulness, values). ACT does not aim to reduce distress, rather its goal is to promote better living or a better quality of life despite distress (Hayes, Strosahl & Wilson, 1999). ACT has been shown to have equal or superior efficacy to CBT with a number of psychological and physical health conditions (A-Tjak et al., 2015; Ruiz, 2012).
  Other Names: Acceptance and Commitment Therapy

SUMMARY:
Title: Acceptance and Commitment Therapy for older adults experiencing psychological distress: A hermeneutic single case efficacy design (HSCED) series.

Anxiety and depression in older age is associated with increased level of disability and lower quality of life (OAs). Unfortunately, pharmacological treatments are disproportionality relied upon to manage the mental health of OAs. Despite cognitive behaviour therapy (CBT) being the recommended psychotherapy, there is evidence that CBT is less effective for OAs than younger populations.

An alternative treatment, Acceptance and Commitment Therapy (ACT), has been shown to be effective in reducing distress for OAs experiencing physical health difficulties. Several case studies have also indicated that ACT can be effective for OAs with psychological difficulties. ACT aims to change how a person interacts with their thoughts/feelings; to reduce avoidance; and to promote value-focused living.

The study aims to use an adjudicated HSCED to answer the following questions:

i) Is ACT an effective intervention for older adult clients experiencing psychological distress.

ii) Do meaningful changes occur for client-participants over the course of ACT intervention?

iii) What specific factors (ACT-specific, non-specific, extra-therapeutic) contribute to observed changes?

iv) Are observed changes broadly attributable to the ACT intervention?

v) What adaptations may facilitate change when using ACT with older adult clients.

For the study, up to four participants will be recruited from an OA community mental health team, each receiving up to 12 individual sessions of ACT. Participants will be required to complete a number of questionnaires throughout the study, including before/after sessions. Post-treatment, there will be a semi-structured 1:1 interview to explore any changes participants experienced, before a six-week follow-up is employed to check stability of change.

DETAILED DESCRIPTION:
This study aims to investigate whether Acceptance and Commitment Therapy (ACT) is an effective psychotherapeutic intervention for older adults experiencing psychological distress; what processes contribute towards psychological change; and what adaptations may be required to optimise ACT for older adults. There is currently an over-reliance on pharmacological treatments to manage older adult mental health (Andreescu & Reynolds, 2011), and a lack of inclusion of older adult in efficacy studies of psychological treatments (Gatz, 2006). Cognitive behaviour therapy (CBT) is the most evidence-based psychological treatment for mental health conditions. It emphasises the link between thoughts and feelings, and uses cognitive restructuring to facilitate improvement in psychological symptoms. However, of the studies that have included older adults, there is evidence that CBT has a lower effect size in older adults than with working age adults (Kishita & Laidlaw, 2017). There are a number of possible reasons for this, including a lack of age specific adaptations, the over focus on diagnosis specific treatment protocols in CBT, and the increasing physical and psychological co-morbidity associated ageing.

ACT is a trans-diagnostic approach which aims to promote better living by supporting clients through six key processes (e.g. mindfulness, values). ACT does not aim to reduce distress, rather its goal is to promote better living or a better quality of life despite distress (Hayes, Strosahl & Wilson, 1999). ACT has been shown to have equal or superior efficacy to CBT with a number of psychological and physical health conditions (A-Tjak et al., 2015; Ruiz, 2012). We propose that ACT would be especially suitable for older adult clients due to the high rate of co-morbidity older adults experience and the reduced ability to change aspects of these.

However, there is a lack of understanding about the processes by which ACT works (Öst, 2014). Randomised controlled trails (RCTs) are the standard research methodology to investigate psychotherapy efficacy. Due to the stringent criteria required for RCT analyses, there is a limit to how transferrable the findings of an RCT can be to clinical populations (i.e. heterogenous groups). As such, a hermeneutic single case efficacy design (HSCED) is an ideal methodology to employ to identify what contributes towards change for each client. HSCED benefits from high ecological validity, whilst actively focusing on non-specific factors (components common to all psychotherapies, e.g., therapeutic alliance) and extra-therapeutic factors (components that are not related to the therapy, usually participant factors) to delineate change processes.

The research proposal has been developed as part of a Doctoral Thesis in Clinical Psychology. This involved various research presentations panels and submission of an initial research protocol. These are designed to guide the decision-making process and gain feedback from the course research team. As part of the doctoral program, each trainee is allocated a Primary and Secondary Research Supervisor (both Clinical Psychologists), who aided in shaping the practicalities of this research proposal. Each project also recruits a Field Supervisor who supports with expertise in the project area. Participants will be recruited from the service the Field Supervisor is employed at, thereby creating a direct level of clinical supervision that is paramount to psychotherapy.

Participants will be informed about the study through a member of their healthcare team. The service will ensure potential participants have the capacity to consent to treatment and will provide them with an overview of the study. Potential participants will be made aware of informed consent; that they do not have to take part and that declining to take part will in no way affect their treatment from the service. If a participant declines to take part at this stage, they will be offered treatment as usual from the service. If they consent to take part, the researcher will contact them the following week to answer any additional questions. This will allow them sufficient time to consider whether they would like to take part or not.

This research aims to use a sample that is representative of older adults presenting with psychological distress. See Inclusion/Exclusion sections for further explanation of these criteria.

This study aims to reflect usual clinical practice where possible; therefore, the burden to participants will be of a similar level to treatment as usual. That is, they will be expected to attend the older adults service for regular one-to-one psychotherapy and to discuss their mental health difficulties, contributing factors and what is maintaining their difficulties. Thus, as with any psychological therapy, there is a potential risk that talking about distressing experiences will cause an increase in frequency or intensity of pre-existing mental health conditions. These risks will be monitored through the study by the Trainee Clinical Psychologist (who is both researcher and therapist) through discussion with the participant, use of outcome measures and importantly by utilising weekly clinical supervision with the Clinical Psychologist at the service. This allows a space for any concerns to be raised and for the service to have clinical oversight of the participants.

The aspects of the study which are additional to usual practice are as follows: participants will be required to complete more questionnaires; and participants will be required to come in for an interview after the block of therapy has ended. Every effort has been made to reduce the burden these place upon participants. For instance, shorter questionnaires have been used where possible. Participants will also be asked about any adaptations required to complete questionnaires (e.g. larger font, someone completing questionnaires with them). Participants will be reimbursed for the aspects of the study which are additional to usual practice.

There are several potential benefits to participants taking part in this research, as suggested by the ACT literature. These include decreased psychological distress, increased psychological flexibility and improved quality of life.

To ensure confidentiality, Participant Study Numbers (PSN) will be assigned to each participant to correspond with treatment data. PSNs will be listed in the Trial Recruitment Log along with participant's name, date of birth and NHS number. All other documents related to the participant will use the PSN only. All researchers will endeavour to protect the rights of the participants to privacy and will adhere to the Data Protection Act, 2018. Only the minimum required information for the purposes of the study will be collected. Participant information will be held securely, in a locked room, or locked cupboard or cabinet. Access to the information will be limited to the study staff and investigators. Computer held data including the study database will be held securely and password protected. All data will be stored on a secure dedicated web server. Access will be restricted by user identifiers and passwords (encrypted using a one-way encryption method). Information about the study in the participant's medical records / hospital notes will be treated confidentially in the same way as all other confidential medical information.

As the main researcher is also the therapist, potential conflict of interests will be managed by: using weekly clinical supervision; fortnightly ACT supervision; a 20% random sampling of the audio recorded sessions to ensure adherence to ACT techniques; and using an independent researcher to carry out the Change Interview. Another benefit of using a HSCED series, is that an independent panel adjudicates on the final outcome as to where change was attributed for each client, reducing the researcher-therapist bias.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 65 years of age.
* Score at least 8 on the Hospital Anxiety and Depression Scale (HADS; ZIgmond & Snaith, 1983) on either the anxiety or depression sub-scale. The HADS is an outcome measure already used by the MHSOP.
* Be referred to the MHSOP for psychological support.
* Have capacity to give informed consent.
* Be willing to engage in one-to-one psychotherapy.
* Be able to travel to the service (either independently or with support).

Exclusion Criteria:

* A score lower than 22-24 on the MoCA. This is to screen for a level of cognitive deficit, which cannot be accommodated for in the current study, due to the adaptations which will be required (e.g. review sessions, carer enrolment to support memory consolidation). Cut-off limit is dependent on the individual's age and education history. The MoCA is administered by the MHSOP as standard practice.
* Not rated higher than Cluster 8 (Mental Health Clustering Booklet 2013/14, Department of Health), a categorisation based on the Health of the Nation Outcome Scale (HoNOS; Wing et al., 1998). Clusters higher than 8 are associated with clients presenting with symptoms of psychosis and it is felt that this level of mental health problem would cause serious heterogeneity between client cases. As standard practice, the MHSOP at Ling Bar Hospital will have rated the client prior to consideration for the study.
* Inability to understand English to a level required to participate fully in the intervention. This is due to a lack of ability to benefit from the intervention without an interpreter, and the impact an interpreter would have on the non-therapeutic processes (e.g. alliance) being measured in this study.
* Not currently undertaking any other psychological therapy, talking therapy or counselling. This is due to the potential impact the other therapy could have on change and the inability to fully account for this.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes — 65 years or older
Enrollment: 3 (Actual)
Dates: Start 2020-04-29 (Actual); Primary Completion 2020-11-18 (Actual); Study Completion 2020-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nima Golijani-Moghaddam, Dr, Principal Investigator — University of Lincoln
Locations (1):
- Mental Health Services for Older People, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Results will be written up in a peer-reviewed journal and as part of a Doctoral Thesis. Individual participant data will be anonymised. Should a request be made for individualised data, this would have to be approved by the various ethical and research boards involved.

REFERENCES:
- [Background] Elliott R. Hermeneutic single-case efficacy design. Psychother Res. 2002 Mar 1;12(1):1-21. doi: 10.1080/713869614. PMID 22471329
- [Background] Hayes SC. Acceptance and commitment therapy: towards a unified model of behavior change. World Psychiatry. 2019 Jun;18(2):226-227. doi: 10.1002/wps.20626. No abstract available. PMID 31059616
- [Background] Ost LG. The efficacy of Acceptance and Commitment Therapy: an updated systematic review and meta-analysis. Behav Res Ther. 2014 Oct;61:105-21. doi: 10.1016/j.brat.2014.07.018. Epub 2014 Aug 19. PMID 25193001
- [Background] A-Tjak JG, Davis ML, Morina N, Powers MB, Smits JA, Emmelkamp PM. A meta-analysis of the efficacy of acceptance and commitment therapy for clinically relevant mental and physical health problems. Psychother Psychosom. 2015;84(1):30-6. doi: 10.1159/000365764. Epub 2014 Dec 24. PMID 25547522
- [Background] Petkus AJ, M A, Wetherell JL. Acceptance and Commitment Therapy with Older Adults: Rationale and Considerations. Cogn Behav Pract. 2013 Feb;20(1):47-56. doi: 10.1016/j.cbpra.2011.07.004. PMID 26997859

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Psychological Therapy
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Psychological Therapy
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.67 (5.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White British | 3
Older People's Quality of Life questionnaire, brief version (OPQOL-brief) [Mean (Standard Deviation); unit: units on a scale] — Older adult specific quality of life measure, based on a longer form version developed from large older adult (mainly non-clinical) cohort study. Scores range from 13-65. Higher scores indicating greater quality of life.
  units on a scale | 43.67 (7.57)
Hospital Anxiety and Depression Scale - Anxiety Subscale(HADS-A) [Mean (Standard Deviation); unit: units on a scale] — Measure of anxiety that is less sensitive to physiological impact, avoiding overlap with physical health conditions. Scores range from 0-21, with higher scores indicating greater anxiety. 8-10 = mild range; 11-15 = moderate; 16+ = severe.
  units on a scale | 13.67 (6.66)
Hospital Anxiety and Depression Scale - Depression Subscale (HADS-D) [Mean (Standard Deviation); unit: units on a scale] — Measure of depression that is less sensitive to physiological impact, avoiding overlap with physical health conditions. Scores range from 0-21, with higher scores indicating greater depression. 8-10 = mild range; 11-15 = moderate; 16+ = severe.
  units on a scale | 9.67 (3.06)
Comprehensive Assessment of Acceptance and Commitment Therapy processes, short-form,(CompACT-8) [Mean (Standard Deviation); unit: units on a scale] — Process outcome measure for acceptance and commitment therapy. Total score indicates level of psychological flexibility the client has. Scores range from 0-48 with greater scores indicating greater psychological flexibility.
  units on a scale | 20 (1.73)

OUTCOME MEASURES:

1. Primary Outcome: Change in Quality of Life Assessed Using the Older People's Quality of Life Questionnaire (OPQOL-brief).
Description: Brief measure of quality of life (QoL) in older age.
Time Frame: up to 20 weeks
Population: All participants completed baseline of 3 or 4 weeks. OPQOL-brief was used at baseline, mid, end, and follow-up point. Missing data was treated as missing. Mean score for all participants at one-month follow-up point shown below.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychological Therapy
Number analyzed (Participants) | 3
score on a scale | 43.33 (8.39)

2. Secondary Outcome: Client's Level of Cognitive Functioning Assessed Using the Montreal Cognitive Assessment (MoCA).
Description: A brief cognitive screening questionnaire which will be administered by the usual care team at the start of the study.
Time Frame: up to 5 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Symptoms of Anxiety and Depression Assessed With the Hospital Anxiety and Depression Scale (HADS).
Description: A brief measure of anxiety and depression that is less prone to conflation of physical health symptoms onto symptoms of psychological distress.
Time Frame: up to 20 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Change in/Progress on Client's Goals Assessed Using the Simplified Personal Questionnaire (PQ).
Description: This consists of up to ten problem statements the client outlines at start of therapy and rates on a 7-point Likert scale for how much they have been bothered by the problem in the past week. They will then re-rate this before each therapy session and again at six-week follow-up.
Time Frame: up to 20 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Change in Client's Weekly Level of Quality of Life Assessed Using the Outcome Rating Scale (ORS).
Description: A brief measure of patient rated outcomes in therapy session.
Time Frame: up to 20 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Change in Therapeutic Alliance Assessed With the Session Rating Scale (SRS).
Description: A brief measure of patient rated therapeutic alliance.
Time Frame: up to 20 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Client's (Qualitative) Views on Individual Therapy Sessions Assessed With the Helpful Aspects of Therapy Form (HAT).
Description: A qualitative measure of patient rated therapeutic alliance.
Time Frame: up to 20 weeks
Reporting Status: Not Posted

8. Secondary Outcome: Change in Psychological Flexibility Assessed Using the CompACT
Description: An ACT process measure.
Time Frame: up to 20 weeks
Reporting Status: Not Posted

9. Secondary Outcome: Client's Attribution of Change and View on Therapy Assessed With the Change Interview
Description: A semi-structured interview to determine the participant's view on any change achieved during therapy. Delivered by a researcher other than the therapist.
Time Frame: up to 20 weeks
Reporting Status: Not Posted

10. Secondary Outcome: Adherence to ACT Related Processes Assessed With the ACT Fidelity Measure (ACT-FM).
Description: A fidelity measure to ensure that sessions meet the requirements of ACT.
Time Frame: up to 20 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Psychological Therapy
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-07): https://cdn.clinicaltrials.gov/large-docs/45/NCT04280445/Prot_SAP_000.pdf